CLINICAL TRIAL: NCT03955796
Title: Capsular Bag Performance of a Hydrophilic and a Hydrophobic Acrylic Intraocular Lens of Similar Design
Brief Title: Performance of a Hydrophilic and a Hydrophobic Intraocular Lens of Similar Design
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes will be made in the design of one of the study IOLs
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ray hydrophobic
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Cataract
Keywords: Cataract, cataract surgery, intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RayOne Hydrophobic Aspheric (Experimental): Patient will receive the hydrophobic IOL during cataract surgery
  Interventions: Device: Hydrophobic IOL
- RayOne Aspheric (Experimental): Patient will receive the non-hydrophobic IOL during cataract surgery
  Interventions: Device: Non-hydrophobic IOL

INTERVENTIONS:
Device: Hydrophobic IOL — RayOne Hydrophobic Aspheric, hydrophobic IOL
  Arms: RayOne Hydrophobic Aspheric
Device: Non-hydrophobic IOL — RayOne Aspheric, non-hydrophobic IOL
  Arms: RayOne Aspheric

SUMMARY:
Comparison of the capsular bag performance of the RayOne Hydrophobic Aspheric with the RayOne Aspheric

DETAILED DESCRIPTION:
Cataract surgery is nowadays considered a safe surgery with a short rehabilitation time for the patients. Two main problems arising post-surgically are the predictability and stability of the implanted intraocular lens (IOL) in the capsular back and the formation of posterior capsule opacification (PCO). The performance of the IOL in the capsular bag influences the anterior chamber depth (ACD), tilt and decentration of the IOL, as well as formation of PCO. The main source of error for calculation of IOL power is an inaccurate prediction of the post-surgical ACD resulting in short- or farsightedness. Furthermore, capsular fibrosis and phimosis can also lead to tilt and decentration of the intraocular lens.

PCO is one of the most frequent long-term complications after cataract surgery, occuring in about 12% after 1 year, in 21% after 3 years, and in 28% after 5 years post-surgically. PCO arises when lens epithelial cells (LECs) migrate and proliferate, growing in between the IOL and the posterior capsule, leading to decreased visual acuity.

Material and design of the IOL may have an effect on the formation of PCO. It is suggested that 360° square edge design and hydrophobic material of the IOL may help in the prevention of PCO.

Hence, the aim of this study is to evaluate the capsular bag performance of monofocal IOLs with different materials but similar design and their influence on PCO formation.

100 eyes of 50 patients will be included into this study. After randomization one eye is implanted with the hydrophilic IOL, whereas the other eye gets the aspherical IOL. Follow-up visits will be 1 - 2 hours and 1 week after the surgery, as well as 6 months, 12 months, and 24 months post-surgically. During this visit a slit lamp examination, measurement of the intraocular pressure, visual acuity assessment, biometrical measurements of the eye, retroillumination photography and analysis of tilt and decentration of the IOL using the purkinjemeter will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age-related bilateral cataract
* Age 21 or older
* Visual acuity > 0.05
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Written informed consent prior to surgery

Exclusion Criteria:

* Relevant other ophthalmic diseases such as pseudoexfoliation syndrome (PEX), Intraoperative Floppy Iris Syndrome (IFIS), cornea pathologies
* Previous ocular surgery or trauma
* Pregnancy (pregnancy test will be taken in women of reproductive age)

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Anterior chamber depth (ACD) | 24 months
  The change in anterior chamber depth (ACD) before and after surgery will be measured using the IOL Master 700 and compared between the two different IOLs

SECONDARY OUTCOMES:
Distance visual acuity | 24 months
  Uncorrected and corrected distance visual acuity will be determined using ETDRS-charts in a distance of 4 meters and differences in refraction will be compared between the two IOLs
Intraocular pressure | 24 months
  Intraocular pressure will be measured before and after surgery using non-contact-tonometry and differences will be compared between the two differen IOLs

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided